CLINICAL TRIAL: NCT02794688
Title: Ductal Lavage in Non-lactating Female Women With Mastitis: A Single Arm, Observational Study
Brief Title: Ductal Lavage in Non-lactating Female Women With Mastitis
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangzhou Jie Jian Instrument Co,Ltd (Unknown); China Anti-aging Promoting Association (Other)
Responsible Party: Principal Investigator, Shunrong Li, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: DLNLM-01
Record Dates: First submitted 2016-05-24; First posted 2016-06-09 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Mastitis
Keywords: Non-lactating; idiopathic granulomatous mastitis; periductal mastitis; ductal lavage
MeSH Terms: conditions — Mastitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All patients are required to have biopsy to exclude breast carcinoma. The storage of the biospecimen will follow the standard of practices of Sun Yat-sen Memorial Hospital.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ductal lavage group: The patients will receive ductal lavage therapy every other day for two weeks, and will be followed up for one year.
  Interventions: Procedure: Ductal lavage therapy

INTERVENTIONS:
Procedure: Ductal lavage therapy — 1. Patient lies in supine position, with routine sterilizing and draping procedure.
  2. Local anesthesia with 2ml lidocaine (1%) around the nipple.
  3. Identification of 4-5 openings of the lactiferous ducts from the nipple.
  4. Insertion of all infusion cannula (21-23G ) into the identified openings of the lactiferous ducts.
  5. Start the infusion pump with 15ml irrigation solution (2% Lidocaine 5ml, Triamcinolone acetonide 40mg，0.9% saline 10ml and ceftriaxone 1.0g). If the patients had elevated white blood cell count and fever (>38 celsius degree), oral intake or infusion of antibiotics were allowed, when necessary.
  6. The patient returns to the clinic the next day, with the irrigation solution staying in the lactiferous ducts overnight, and receives breast massage.
  7. Repeat step 1-6 every other day for 2 weeks.
  8. Fine needle aspiration is allowed. Oral intake of corticosteroids, excisional drainage or surgery are not allowed.

SUMMARY:
RATIONALE and PURPOSE: For non-lactational mastitis patients pathologically diagnosis of idiopathic granulomatous mastitis (IGM) or periductal mastitis (PD), the investigators hypothesized that ductal lavage is able to relieve the symptoms and achieve complete response, with shorter recovery time than oral intake of antibiotics or corticosteroids treatments. This single arm, observational, case series, pilot study is going to evaluate the effectiveness of ductal lavage in patients with non-lactational IGM or PD.

DETAILED DESCRIPTION:
Inflammatory non-lactating breasts diseases encompasses a large spectrum of diseases ranging from infective diseases to autoimmune diseases, which cause considerable morbidity and difficulty in diagnosis. In daily practices, exclusion of possible diagnosis of breast carcinoma is the most important step. Aetiological factors for non-lactational mastitis include bacterial infection, tuberculosis, auto-immune disorders, etc. Treatments for these patients including antibiotics, anti-tuberculosis therapy, and corticosteroids treatments. Many of these patients were pathologically diagnosed as periductal mastitis (PD) or idiopathic granulomatous mastitis (IGM). The current treatment for PD or IGM include corticosteroids treatments, antibiotics and surgical treatments. Based on literature review, the complete response (CR) rate of corticosteroids and surgical treatment ranged between 63-87% and 89-100%, respectively. Time to CR ranged between 2-8 month for corticosteroid treatment.

Pathological findings of patients of IGM or PD revealed infiltrating inflammatory cells and neutrophilic microabscesses around the lobular units and partial ductal obstruction, we hypothesized that ductal lavage therapy will be able to relieve the symptom by dilating the lactiferous duct followed by irrigation solution flushing, with shorter recovery time and satisfactory CR rate. In our institution(Sun Yat-sen Memorial Hospital,Guangzhou, Guangdong, P.R.China), it is our routine practice to perform ductal lavage therapy to patients with non-lactating breasts diseases, especially for patients with IGM or PD, before we start corticosteroid or antibiotics treatments. For patients with evidence of bacterial infection, antibiotics was added into the irrigation solution. In our experience, many patients had short recovery time and low relapse rate, sparing the use of corticosteroid or antibiotics treatments. However, there is no concrete data to quantify the efficacy of ductal lavage therapy for IGM or PD patients. This observational study aims to prospectively enroll eligible patients and investigate the efficacy of ducal lavage therapy in IGM or PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Female, age between 18 and 65 years old.
* Inform consent signed.
* Clinical diagnosis of non-lactating mastitis, defined as mastitis occurred more than 1 year after the cessation of lactation.
* Never receive any treatments after the cessation of lactation.
* Good health, judged by clinicians, to receive ductal lavage.
* Pathologically diagnosed as idiopathic granulomatous mastitis (IGM) or periductal mastitis (PD).

Exclusion Criteria:

* Pathological diagnosis of breast carcinoma.
* Pregnant women.
* Evidences suggest possible diagnosis of systemic lupus erythematosus(SLE), rheumatic disorders or other systematic auto-immune diseases.
* Evidences suggest possible diagnosis of tuberculosis.
* Imaging examinations indicates foreign objects retained in the breast
* Evidences suggest possible diagnosis of fungus infection of the breast
* Patients with inappropriate coagulation function, cardiac function, pulmonary function, liver and renal function, that clinicians judges as not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with non-lactating mastitis, pathologically diagnosed as idiopathic granulomatous mastitis (IGM) or periductal mastitis (PD), were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Time to complete response | Time from the initial treatment to first assessment of complete response, reported between day of first treatment and 1 year thereafter.
  The length of time from the date of initial treatment to the date of complete response. Complete response (CR) was defined as reaching all of the followings: 1) visual analogue score <=1; 2) Disappearance of all local symptoms, such as redness, pain, swollen, etc. 3) Disappearance of fistula, if any; 4) The patient can return to normal life without any medical assistant.5) Disappearance of palpable or ultrasound detectable mass were defined as physical-CR and imaging-CR, respectively.

SECONDARY OUTCOMES:
Complete response rate | Evaluations were performed every week for the 1st month, and every other month thereafter until complete response, reported between the day of first treatment and 1 year thereafter.
  The proportion of patients with complete response within 1 year after the initial treatment.
Partial response rate | Evaluations were performed every week for the 1st month, and every other month thereafter until partial response, reported between the day of first treatment and 1 year thereafter.
  The proportion of patients with partial response within 1 year after the initial treatment. Partial response was defined as reaching all of the followings: 1) decreased visual analogue score>=2; 2) Significantly relieved of all local symptoms, such as redness, pain, swollen, etc. 3) Disappearance of spontaneous discharge through fistula, if any; 4) The patient stated that the symptom is relieved significantly.5) Size of the target mass (Largest dimension) is reduced >30%, compared with that of the baseline. Partial response assessed by physical and ultrasound were defined as physical-partial-response and imaging-partial-response, respectively.
Relapse incidence after complete response | Evaluations were performed every week for the 1st month, and every other month thereafter until relapse, reported between the day of complete response and 1 year after the initial treatment.
  The incidence of relapse after complete response, within 1 year after the initial treatment. Definition of relapse including any of the followings: 1) Notice of new palpable mass; 2) Notice of new fistula; 3) Notice of new local symptoms, such as pain, redness, swollen and heated skin. Only patients with complete response during the study follow-up will be assessed for this outcome.
Progression incidence after partial response | Evaluations were performed every week for the 1st month, and every other month thereafter until disease progression, reported between the day of partial response and 1 year after the initial treatment.
  The incidence of progression after partial response, within 1 year after the initial treatment. Definition of progression including any of the followings: 1) Progression of local symptoms (redness, swelling, tenderness, pain, fever) significantly. ; 2) Notice of new fistula; 3) The size of the target mass (Largest dimension) increased >20%, compared with that of the day of partial response. Only patients with partial response during the study follow-up will be assessed for this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shunrong Li, M.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Erwei Song, M.D., Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun-Yat-Sen Memorial Hospital of Sun-Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (de-identified) is available upon request.

REFERENCES:
- [Background] Bouton ME, Jayaram L, O'Neill PJ, Hsu CH, Komenaka IK. Management of idiopathic granulomatous mastitis with observation. Am J Surg. 2015 Aug;210(2):258-62. doi: 10.1016/j.amjsurg.2014.08.044. Epub 2015 Feb 7. PMID 25746911
- [Background] Gautier N, Lalonde L, Tran-Thanh D, El Khoury M, David J, Labelle M, Patocskai E, Trop I. Chronic granulomatous mastitis: Imaging, pathology and management. Eur J Radiol. 2013 Apr;82(4):e165-75. doi: 10.1016/j.ejrad.2012.11.010. Epub 2012 Nov 29. PMID 23200627
- [Background] Gopalakrishnan Nair C, Hiran, Jacob P, Menon RR, Misha. Inflammatory diseases of the non-lactating female breasts. Int J Surg. 2015 Jan;13:8-11. doi: 10.1016/j.ijsu.2014.11.022. Epub 2014 Nov 22. PMID 25447605
- [Background] Lacambra M, Thai TA, Lam CC, Yu AM, Pham HT, Tran PV, Law BK, Van Nguyen T, Pham DX, Tse GM. Granulomatous mastitis: the histological differentials. J Clin Pathol. 2011 May;64(5):405-11. doi: 10.1136/jcp.2011.089565. Epub 2011 Mar 8. PMID 21385894
- [Derived] Chen K, Zhu L, Hu T, Tan C, Zhang J, Zeng M, Li S, Song E. Ductal Lavage for Patients With Nonlactational Mastitis: A Single-Arm, Proof-of-Concept Trial. J Surg Res. 2019 Mar;235:440-446. doi: 10.1016/j.jss.2018.10.023. Epub 2018 Nov 19. PMID 30691827